CLINICAL TRIAL: NCT07207967
Title: End-Inspiratory Pause Enhances Ventilation Efficiency Without Affecting autoPEEP in COPD Patients During Controlled Ventilation
Brief Title: End-Inspiratory Pause in COPD Patients During Controlled Ventilation
Acronym: PYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, Joaquin Pérez, Sanatorio Anchorena San Martin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10/2024
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: mechanical ventilation; COPD; End-inspiratory pause; AutoPEEP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO PAUSE ventilation (Active Comparator): Patients will be ventilated in volume-controlled mode with square-flow waveform, without end-inspiratory pause, tidal volume of predicted body weight (VtPBW) 6-8 ml/kg, TI 0.6-0.8 seconds, RR 10-16 breaths per minute (bpm) and I:E relationship 1:4-1:8. External positive end-expiratory pressure (PEEPext) will be set to the maximum value that did not increase plateau pressure (Pplat) ≥ 1cmH2O compared to zero PEEP, and FiO2 to maintain oxygen saturation of 90-95%.
  Interventions: Other: NO PAUSE VENTILATION
- PAUSE ventilation (Experimental): Patients will be ventilated in volume-controlled mode with square-flow waveform, where total Ti will be the same that during NO PAUSE ventilation, but inspiratory flow will be increased and a part of the total inspiratory time will be replaced by end-inspiratory pause of 0.3-0.5 s. All the remaining parameters will be equal to the NO PAUSE ventilation phase. Tidal volume of predicted body weight (VtPBW) 6-8 ml/kg, TI 0.6-0.8 seconds, RR 10-16 breaths per minute (bpm) and I:E relationship 1:4-1:8. External positive end-expiratory pressure (PEEPext) will be set to the maximum value that did not increase plateau pressure (Pplat) ≥ 1cmH2O compared to zero PEEP, and FiO2 to maintain oxygen saturation of 90-95%.
  Interventions: Other: END INSPIRATORY PAUSE DURING CONTROLLED VENTILATION

INTERVENTIONS:
Other: END INSPIRATORY PAUSE DURING CONTROLLED VENTILATION — PATIENTS WILL BE VENTILATED WITH END-INSPIRATORY PAUSE AND HIGH INSPIRATORY FLOW DURING CONTROLED VENTILATION
  Arms: PAUSE ventilation
Other: NO PAUSE VENTILATION — PATIENTS WILL BE VENTILATED IN VOLUME CONTROLLED VENTILATION WITHOUT END-INSPIRATORY PAUSE
  Arms: NO PAUSE ventilation

SUMMARY:
In patients with airflow obstruction receiving mechanical ventilation, an important objective is to reduce lung hyperinflation often using controlled hypoventilation[1]. At the same time, maintaining acceptable gas exchange is challenging, as major reductions in minute ventilation (VE) raises carbon dioxide (CO2) and causes respiratory acidosis, which may lead to adverse physiological consequences.

Relatively prolonged end-inspiratory pause (EIP) has been shown to optimize CO2 clearance in hypoxemic mechanically ventilated patients[2]. Previous data suggests that, at equivalent total inspiratory-time (TI), shorter insufflations followed by EIP can enhance CO2 elimination in acute lung injury [3]. Adding EIP is classically discouraged in chronic obstructive pulmonary disease (COPD) because - at constant respiratory rate (RR) - prolonging inspiration reduces expiratory time (TE), and can worsen hyperinflation and impair hemodynamics[4, 5].

In this study, we assessed whether a breathing pattern characterized by high inspiratory flow (V ̇) plus EIP could reduce PaCO2 without inducing hyperinflation, compared with same inspiration-to-expiration time (I:E) and a ventilation pattern without EIP in patients with COPD undergoing controlled hypoventilation.

Methods We performed a prospective, single-center, cross-over, randomized trial (ethical approval #10/2024) including deeply sedated and intubated adults with COPD exacerbation, PaCO2 ≥ 45 mmHg and no signs of respiratory effort. Persistent air-leaks, severe hemodynamic instability, pregnancy or intracranial hypertension were exclusion criteria. Patient's next of kin signed the informed consent.

At inclusion, we collected demographic characteristics and baseline respiratory variables. A CT-emphysema score[6], using computed tomographies obtained within 24 hs of intubation for clinical reasons, was calculated (A.R, a pulmonologist specialized in medical imaging). Each lung was divided into 3 regions (superior, medium and inferior) based on anatomical references and were graded as no emphysema (score 0), emphysema ≤25% (score 1), ≤50% (score 2), ≤75% (score 3) and >75% (score 4). Scores of the six regions were summed to obtain the total score, giving a minimum 0 and a maximum of 24 points. Total scores ≥ 2 are indicative of emphysema.

Patients were ventilated in volume-controlled mode with square-flow waveform, tidal volume of predicted body weight (VtPBW) 6-8 ml/kg, TI 0.6-0.8 seconds, RR 10-16 breaths per minute (bpm) and I:E relationship 1:4-1:8. External positive end-expiratory pressure (PEEPext) was set to the maximum value that did not increase plateau pressure (Pplat) ≥ 1cmH2O compared to zero PEEP[7], and FiO2 to maintain oxygen saturation of 90-95%.

Two ventilation strategies, each one applied for 30 minutes, were randomly evaluated (Figure 1A): a) ventilation without EIP, using initial ventilator settings (VentNO-PAUSE); b) ventilation with EIP (VentPAUSE), in which V ̇ was increased and 40-50% of the total inspiratory time (TI) was replaced by EIP; the remaining setting were equal to VentNO-PAUSE. At the end of each phase, we collected arterial blood gases, respiratory mechanics and basic hemodynamics. Total PEEP (i.e., PEEPtot=PEEPext + autoPEEP) and Pplat were assessed with 5-second end-expiratory, and 2-second end-inspiratory occlusions, respectively. Driving airway pressure (ΔP) was computed as Pplat - PEEPtot, normalized elastance (ERS-n) as driving pressure (ΔP)/VtPBW and inspiratory airway resistance (Raw) as (Peak pressure [Ppeak] - Pplat) / V ̇.

We hypothesized that ventilation efficiency would be better during VentPAUSE, and wanted to evaluate whether this strategy would have allowed to reduce VE while keeping the same CO2 obtained without EIP. Accordingly, and assuming a constant CO2 production, we calculated the predicted VE during VentPAUSE to maintain the same CO2 measured during VentNO-PAUSE with the formula :

Predicted VE_( (Vent_PAUSE))=█(〖PaCO_(2 )〗_((Vent_PAUSE ) )@ )/〖PaCO_2〗_((Vent_(NO-PAUSE) ) ) × VE used during the study phases [8] This allowed to calculate to what extent it would have been possible to reduce VE (VEpred) and RR (RRpred) using the experimental strategy. We additionally calculated the predicted prolongation of expiration using the new RRpred as: TE-pred = (60/RRpred) - TI.

We calculated the ventilatory ratio as an indice reflecting physiological dead-space ventilation (VD/VT)[9].

ELIGIBILITY:
Inclusion Criteria:

* deeply sedated and intubated adults with COPD exacerbation, PaCO2 ≥ 45 mmHg and no signs of respiratory effort
* sign the informed consent

Exclusion Criteria:

* Persistent air-leaks, severe hemodynamic instability, pregnancy or intracranial hypertension were exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Arterial pressure of carbon dioxide | 30 min
  Arterial pressure of carbon dioxide
arterial pH | 30 min
  arterial pH

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena San Martín, San Martín, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
confidential data